CLINICAL TRIAL: NCT04712968
Title: Efficacy of Daylight as Adjunctive Treatment in Patients With Unipolar Depression - a Randomized Controlled Feasibility Study
Brief Title: Efficacy of Daylight as Adjunctive Treatment in Patients With Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis of preliminary results indicated a need for protocol re-design.
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aarhus universitet
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2021-09

CONDITIONS: Unipolar Depression
Keywords: Dayligt; Major Depression; Light Therapy; Sleep; Unipolar depression; Adjunctive treatment; Circadian rhythm
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (intervention group) (Experimental): Regular exposure to morning daylight
  Interventions: Behavioral: Regular exposure to morning daylight
- Group 2 (control group) (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: Regular exposure to morning daylight — Participants are asked to stay outside in morning daylight for minimum 30 minutes each day before 1 pm for 6 weeks. A specific plan for individual outdoor possibilities for daylight exposure is made (e.g. a walk, a stay in a park or in their garden, a bike trip). Furthermore a detailed instruction to the personal light tracker "LYS Button" and the matching "LYS Insight app" is provided. The "LYS Insight app" gives the user access to real-time insight of light stimulus. Further, the participants receive psycho-education on the connection between exposure to morning daylight and antidepressant effect. All participants in this group receive the intervention as add-on to usual treatment, which may comprise prescribed antidepressants, psychotherapy, including psycho-education and psychiatric care.
  Arms: Group 1 (intervention group)

SUMMARY:
The aim of this study is to improve the treatment effect for outpatients with depression by adding regular daily morning daylight exposure to their treatment with antidepressants. Patients will wear a personal light tracker to keep them motivated. Our hypothesis is that patients daily exposed to morning daylight, as a supplement to standard treatment for depression, will achieve significantly higher antidepressant effect that patients receiving standard treatment alone. Furthermore, we hypothesize that they will experience improved well-being and sleep.

DETAILED DESCRIPTION:
Due to inadequate efficiency of existing medical and psychotherapeutic treatments for depression there is a need for investigating the efficacy of adjunctive treatments. Light therapy has proven efficient as an add-on treatment for depression, but some patients might prefer being outdoors rather than sitting in front of a light therapy screen. However, no high-quality studies, have so far investigated the antidepressant and other potential positive effects of regular exposure to morning daylight for patients with unipolar depression.

The aim of this study is to examine the efficacy of morning daylight as add-on to treatment as usual in patients with depression. Efficacy is measured as reduction of depressive symptoms, improvement of sleep quality, and improvement of well-being.

Methods and material: A randomized controlled trial comprising 150 patients diagnosed with unipolar depression aged 18-50 years will be conducted. Patients are included after giving informed consent and the study period is 6 weeks. A wearable Personal Light Tracker, measuring the amount off light received, will be provided for all participants. Participants will be randomized into the following groups:

Group 1: Daylight (outdoor daylight exposed stay for minimum 30 minutes per day before 1 pm). To motivate patients to go outside they will receive psychoeducation on the connection between exposure to morning daylight and a possible antidepressant effect, and they are introduced to potential options for outdoor activities. A detailed instruction to the personal light tracker and the matching app, for monitoring the amount of light received throughout the day, is provided.

Group 2: Control group receiving treatment as usual. Patients will wear a personal light tracker but they are not introduced to the light-monitoring-app.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling criteria for an ICD-10 diagnosis of unipolar depression (F. 32.0, F.32.1, F.32.2, F32.3, F. 32.8. F.33.0, F.33.1, F.33.2, F. 33.3)
* Hamilton Depression Score (HAM-D17) ≥ 12
* In treatment with the same antidepressant medication 14 days prior to inclusion
* The participant must have access to a smart phone

Exclusion Criteria:

* Actual treatment with Electro Convulsive Therapy (ECT)
* Seasonal Affective Disorder (SAD)
* Known sleep disturbances (sleep-apnoea, narcolepsy, or "restless legs syndrome")
* On lithium, agomelatine, melatonin and/or mirtazapine
* Known eye disorders
* Current alcohol- or drug abuse
* Current user of Light therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | Is measured at inclusion (baseline/ week 0), at week 2 and at week 6 (endpoint).
  Measured on the Hamilton Depression Rating Scale interviewbased 17 item version (HAM-D17).The scale ranges from 0 to 52; the higher the score the more depressed is the patient.
Change in depressive symptoms | Participants will answer the questionnaire every fourth day in the 42 day studyperiod.
  Measured on Hamilton Depression Scale: selfreported version (HAM-D6). A questionnaire measuring depressive symptoms. The scale ranges from 0-22, the higher the score the more depressed is the patient.
Change in sleep quality | Is measured at inclusion (baseline/ week 0) and at week 6 (endpoint).
  Measured by Pittsburgh Sleeping Quality Index (PSQI).The score is between 0 and 21 "0" indicating no difficulty and "21" indicating severe difficulties.
Change in insomnia severity | Is measured at inclusion (baseline/ week 0), at week 2 and at week 6 (endpoint).
  Measured by Insomnia Severity Index (ISI). Self-report instrument measuring the patient's perception of insomnia. The scale ranges from 0 to 28. The higher the score the more severe insomnia.
Change in well-being | Is measured at inclusion (baseline/ week 0), at week 2 and at week 6 (endpoint).
  Measured on The WHO-5 Well-Being Index (WHO-5). A questionnaire which measures well-being. The scale ranges from 0 to 100, the higher the score the more well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Kragh, PhD, Principal Investigator — Department of Affective Disorders Arhus, University Hospital. Psychiatry
Locations (1):
- "Psykiatriens Hus" Department of Affective Disorders Arhus, University Hospital. Psychiatry, Aarhus, Denmark